CLINICAL TRIAL: NCT07111052
Title: Lock and Protect: An Emergency Department Randomized Controlled Trial to Reduce Adolescent Access to Lethal Means of Suicide
Brief Title: Lock and Protect: Reducing Adolescent Access to Lethal Means of Suicide
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: Columbia University (Other)
Responsible Party: Principal Investigator, Ashley Blanchard, Assistant Professor of Pediatrics in Emergency Medicine, Columbia University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: AAAV6627
Record Dates: First submitted 2025-08-06; First posted 2025-08-08 (Actual); Last update posted 2025-12-05 (Actual); Status verified 2025-12

CONDITIONS: Suicide; Suicide Attempt; Adolescent Suicidality; Suicide Ideation
Keywords: adolescent suicide; lethal means counseling; lethal means access; adolescent suicide prevention
MeSH Terms: conditions — Suicide; Suicide, Attempted

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Lock and Protect, web-based lethal means counseling intervention (Experimental): Guardians and patients will receive the intervention, Lock and Protect, is a user-friendly web-based decision aid that identifies preferences and explores options for removing or storing lethal means safety.
  Interventions: Behavioral: Lock and Protect is a self-administered, web-based decision aid for caregivers of adolescents at risk for suicide.
- Usual care (No Intervention): All patients enrolled in the study, as part of usual care, will receive evaluation by the pediatric psychiatry team. This includes in-depth interviews about suicide risk and self-harm. All patients enrolled in this study are 1) evaluated by the pediatric psychiatry team and 2) evaluated for safety and suicide risk that informs if inpatient behavioral health admission is warranted based on the assessment. All patients who are eligible for study enrollment, as part of usual care for patients presenting for suicidal thoughts and behaviors or self-harm, will receive standard safety procedures while undergoing evaluation in the ED. These ED specific safety procedures include clinical observation of the patient while deemed to be at risk for any form of self-harm, removal of any phones and/or personal items that may be used for self-harm, being placed in behavioral health specific ED evaluation rooms, and (when warranted) security team presence.

INTERVENTIONS:
Behavioral: Lock and Protect is a self-administered, web-based decision aid for caregivers of adolescents at risk for suicide. — Lock and Protect is a user-friendly web-based decision aid that identifies preferences and explores options for removing or storing lethal means safety through: (a) education on home means of suicide, such as firearms, medications, and other potentially dangerous home and external items/situations (e.g., poisons, methods/ligatures used in suffocation/hanging), and community hazards (e.g., subways, heights); (b) safe storage options; and (c) protective monitoring and supervision as a means of increasing adolescent safety during a time of elevated risk.
  Arms: Lock and Protect, web-based lethal means counseling intervention

SUMMARY:
The primary goal is to determine the acceptability and feasibility of implementing the Lock and Protect decision aid. The secondary goals are to identify the potential short-term impact of Lock and Protect on home firearm and medication storage, parental self-efficacy. Using interviews with caregivers, the study will clarify the acceptability, feasibility, and barriers to implementing the Lock and Protect hone safety plan. This will allow further development of effective strategies to subsequently further test and use Lock and Protect in the ED.

NOTE: The study will only recruit guardians and their adolescents from the pediatric ED at Morgan Stanley Children's Hospital NY-Presbyterian.

DETAILED DESCRIPTION:
Suicide is the second leading cause of death in adolescents in the United States. Suicide rates increased 22% from 2005-2015, with a 28% increase in New York State. Emergency Departments (EDs) capture a medically underserved population at high risk for suicide and provide an important but typically missed opportunity for adolescent suicide prevention. Reducing access to guns, medications, and other methods of suicide (also called lethal means restriction or counseling) is one of the few suicide prevention interventions found to decrease suicides. It is based on the idea that reducing access to highly lethal means of suicide during a time of vulnerability can prevent suicide by decreasing the lethality of attempts. This is of critical importance in adolescence, when the transition from thinking about suicide to committing or attempting suicide is often sudden and unplanned, using the most readily available method to attempt suicide. However, effective tools to facilitate suicide prevention, particularly restricting lethal mean access, are lacking. Our expert team has developed a novel, low-resource, tablet-based intervention termed Lock and Protect intended to decrease risk of suicide in adolescents evaluated in EDs.

The investigator will conduct a research study of parents or caregivers (hereafter referred to as caregivers) who receive the intervention during evaluation of their adolescent in the ED for suicidal ideation, self-ham, or suicide. The study will randomly assign caregivers; those who are assigned to the intervention will receive usual ED care and receive the Lock and Protect intervention. Guardians randomly assigned to receive usual ED care alone will complete study surveys in addition to usual ED care. Usual ED care for patients presenting with self-harm or suicidal thoughts and behaviors includes evaluation by the child psychiatry team and determination of risk to determine if safety planning (Stanley Brown safety plan completed in the medical chart), discharge home, or inpatient psychiatric admission is warranted. The study will enroll parents of youths 13-17 years-old presenting to the ED for suicidal thoughts or behaviors. Caregivers will not be part of the study if their child is medically unstable, a caregiver does not speak English or Spanish, and/or they do not reside in the same home as the patient. The investigator hopes to determine if home access to high-risk medications and/or firearms has changed at 1-month after ED visit. The study will also measure decision quality and behavioral intent through surveys.

ELIGIBILITY:
Inclusion Criteria: (Both caregiver and patient must agree to participation to be eligible)

* Parents or caregivers of adolescents aged 13-17 years presenting to the ED for suicidal thoughts and/or behaviors or non-suicidal self-injury as defined by presenting complaint or initial provider assessment.
* Patients ages 13-17 years-old presenting to the ED for non-suicidal self-injury (NSSI), suicidal thoughts and behaviors

Exclusion Criteria:

* Medically unstable children
* Patients with autism, intellectual disability, or active psychosis
* Lack of parental and/or youth English and/or Spanish fluency
* Caregivers who do not reside in the same home as the patient for at least 2 nights a week
* If the caregiver OR patient does not agree to participation both participants will be excluded

Ages: 13 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 50 (Estimated)
Dates: Start 2025-09-11 (Actual); Primary Completion 2026-12-31 (Estimated); Study Completion 2027-03 (Estimated)

PRIMARY OUTCOMES:
Proportion of caregivers who improved home storage of medications and/or firearms | Baseline (ED visit), 1 month follow-up
  The primary efficacy outcome is change in home access to medications and/or firearms by 1-month post-discharge from the ED, as measured by a REDCap self-administered survey.

SECONDARY OUTCOMES:
Mean Decision Conflict Scale Score (low literacy) | Baseline (ED visit)
  This outcome is designed to measure decision quality. Decision quality is a fundamental element of the Ottawa Decision Support Framework, as a marker of readiness to change. Scores range from 0 (no decisional conflict) to 100 (extremely high decisional conflict).
Number of subsequent ED visits for suicide-related events | From ED enrollment to 3-months after baseline ED visit
  The study will assess subsequent adolescent ED visits for NSSI, suicidal ideation, or suicide attempt, within 3 months of baseline ED visit.
Feasibility of Intervention Measure - Instrument Score | Baseline (ED visit)
  This is to measure feasibility of intervention. A 4-item instrument measuring the feasibility of an intervention. Reported by caregivers, assigned to the intervention arm, after completion of the Lock and Protect intervention.
  Score response range 1-5. Completely disagree (1) Disagree (2) Neither agree nor disagree (3) Agree (4) Completely agree (5)
  Scale is created by averaging the 4 responses.
Acceptability of Intervention: Instrument score | Baseline (ED visit)
  This is to measure acceptability of intervention. A 4-item instrument measuring the acceptability of an intervention. Completed by caregivers assigned to the intervention, after completing the Lock and Protect intervention.
  Score response range 1-5. Completely disagree (1) Disagree (2) Neither agree nor disagree (3) Agree (4) Completely agree (5)
  Scale is created by averaging the 4 responses.

CONTACTS AND LOCATIONS:
Overall Officials: Ashley Blanchard, MD, MS, Principal Investigator — Columbia University
Locations (1):
- Morgan Stanley Children's Hospital, Pediatric Emergency, New York, New York, United States

IPD SHARING:
Plan to Share IPD: Undecided